CLINICAL TRIAL: NCT02910388
Title: Direct Colposcopic Vision and Large Loop Excision of the Transformation Zone in Women With Cervical Dysplasia: a Randomized Controlled Trial.
Brief Title: LLETZ Under Direct Colposcopic Vision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zydolab - Institute of Cytology and Immune Cytochemistry (Other)
Collaborators: Ruhr University of Bochum (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CONE-3
Record Dates: First submitted 2016-09-15; First posted 2016-09-22 (Estimated); Last update posted 2020-06-02 (Actual); Status verified 2017-12

CONDITIONS: Uterine Cervical Dysplasia
Keywords: conization; LLETZ; loop excision; randomized controlled trial; colposcopy; direct colposcopic vision; intraoperative colposcopy
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Colposcopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- LLETZ with colposcopy (Experimental): The LLETZ procedure will be performed under direct colposcopic vision
  Interventions: Device: LLETZ with colposcopy
- LLETZ without colposcopy (Active Comparator): The LLETZ procedure will be performed without colposcopy
  Interventions: Other: LLETZ without colposcopy

INTERVENTIONS:
Device: LLETZ with colposcopy — Loop procedure using a colposcope in order to see and remove the abnormal cervical tissue
  Arms: LLETZ with colposcopy
Other: LLETZ without colposcopy — Loop procedure without using a colposcope
  Arms: LLETZ without colposcopy

SUMMARY:
To assess the benefits of large Loop excision of the transformation Zone (LLETZ) under direct colposcopic Vision.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven cervical dysplasia
* colposcopy Prior to conization
* informed consent

Exclusion Criteria:

* significant language barrier
* a personal history of conization
* pregnancy
* the use of blood thinner
* unwillingness to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
the resected cone mass | 10 minutes
  the resected cone mass will be quantified by weighing the removed tissue with a precision scale located in the operating room

SECONDARY OUTCOMES:
Margin status | 2 Days after conization
  Resection margin is judge as "R0" if abnormal cells are not found in the margin of the biopsy or "R1" if abnormal cells remain in the margin of the biopsy. The histopathological examination will be done by an Independent pathologist
Operation time | 20 minutes
  the time from the beginning of the Operation (start of the electrosurgical method) until the end of the operation (the end of hemostatic interventions) will be measured in minutes
Operative complications | 14 days
  Operative complications defined as necessity to intervene therapeutically up to 14 days postoperatively
number of fragments of the surgical specimen | 10 minutes
  surgeons will count the number of the surgical specimen (1 vs. >1)
the dimensions of the surgical specimens | 2 Days after conization
  The circumference, length and thickness of The surgical specimens will be measured
handling of the device | 30 minutes
  surgeons will score their preference regarding the surgical method using an 11-step visual analogue scale (VAS) for ,(ranging from 0 (,very easy') to 10 (,very difficult')
satisfaction with the device | 30 minutes
  surgeons will score their preference regarding the surgical method using an 11-step visual analogue scale (VAS) for ,satisfaction with the device' (ranging from 0 (,very satisfied') to 10 (,absolutely not satisfied')
Time to complete intraoperative hemostasis | 120 seconds
  the time until complete hemostasis as judged by the surgeon has been achieved, will be measured in seconds
Intraoperative blood loss | 5 hours
  intraoperative blood loss will be measured using the difference in serum hemoglobin one day prior to surgery and within 5 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Ziad Hilal, M.D., Principal Investigator — Zydolab - Institute of Cytology and Immune Cytochemistry
Locations (1):
- Department of Obstetrics and Gynecology of the Ruhr University Bochum, Herne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No